CLINICAL TRIAL: NCT02428881
Title: Open Label Pilot Study to Treat Women With Chronic Urinary Retention or Voiding Dysfunction Due to a Primary Disorder of Sphincter Relaxation (Fowler's Syndrome) With Outpatient Urethral Injections of Botulinum Toxin A (BoNT-A)
Brief Title: Botulinum Toxin A Injections in Patients With Fowler's Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08/0216
Record Dates: First submitted 2015-04-08; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Urinary Retention; Fowler's Syndrome
Keywords: onabotulinumtoxin A
MeSH Terms: conditions — Urinary Retention; Fowler Christmas Chapple syndrome | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complete retention- onabotulinumtoxinA (Experimental): Women in complete urinary retention receiving onabotulinumtoxinA
  Interventions: Drug: onabotulinumtoxinA
- Obstructed voiding- onabotulinumtoxinA (Experimental): Women with obstructed voiding receiving onabotulinumtoxinA
  Interventions: Drug: onabotulinumtoxinA

INTERVENTIONS:
Drug: onabotulinumtoxinA — Patients received 100U onabotulinumtoxinA injection into the external urethral sphincter
  Other Names: Botox

SUMMARY:
Hypothesis / aims of study

Urinary retention is uncommon in young women, and one cause is a primary disorder of urethral sphincter relaxation, characterised by an elevated urethral pressure profile and specific findings in the urethral sphincter EMG (Fowler's Syndrome). Women may present with symptoms of obstructed voiding or complete urinary retention. Clean intermittent self-catheterisation is often painful to perform and currently, the only treatment to show benefit is sacral neuromodulation. This aim of this pilot study is to assess the efficacy of urethral sphincter injections of botulinum toxin, defined as improvement of flow rates by more than 50%, improvement in residual volume and scores on the IPSS questionnaire, and safety, in women with Fowler's Syndrome.

Study design, materials and methods In this open label pilot institutional review board approved study, ten women with a primary disorder of urethral sphincter relaxation (elevated urethral pressure profile (UPP), sphincter volume and abnormal EMG) presenting with obstructed voiding (n=5) or in complete urinary retention (n=5) are recruited from a single tertiary referral centre. Baseline symptoms are being assessed using the IPSS questionnaire, and urinary flow and post-void residual volume were measured. After 2% lidocaine injection, 100U of onabotulinumtoxintypeA is being injected into the striated urethral sphincter, divided on either side, under EMG guidance. Patients are being reviewed at weeks 1, 4 and 10 post-treatment and symptoms are reassessed using the IPSS questionnaire, and urinary flow and post-void residual volume are being measured. The UPP is being repeated at week 4.

DETAILED DESCRIPTION:
Full Title: Open label pilot study to treat women with chronic urinary retention or voiding dysfunction due to a primary disorder of sphincter relaxation (Fowler's syndrome) with outpatient urethral injections of botulinum toxin A (BoNT-A).

Short Title: Botulinum toxin A injections in patients with Fowler's Syndrome Rationale: The department of Uro-Neurology at the National Hospital for Neurology and Neurosurgery attracts approximately 300 new female patients with urinary retention referred from all over the UK a year. A retrospective study showed the commonest diagnosis was a primary abnormality of the striated urethral sphincter or Fowler's syndrome. Fowler's syndrome (FS) is due to an intrinsic muscle disorder causing the muscle to be in a state of constant contraction and is recognized by needle electromyography (EMG) of the striated muscle. In the original description the EMG abnormality was frequently observed in women with clinical features of polycystic ovaries, leading to the hypothesis that the electromyographic abnormality was a consequence of a hormonal abnormality, since it is known that the female urinary sphincter is hormonally dependent. The ongoing abnormal EMG activity is thought to lead to a sustained and involuntary contraction of the sphincter that has a secondary effect of inhibiting detrusor contraction.

A diagnosis of FS is made by finding the characteristic abnormal activity on EMG recording but the findings of an abnormally raised urethral pressure profile and an enlargement of the striated urethral sphincter muscle on ultrasound have been shown to be additional valuable investigations. The only treatment found so far to restore voiding is sacral neuromodulation. This is an expensive, resource intensive surgical intervention, subject to a high revision rate (53%). An alternative management option would be welcomed both by patients and healthcare professionals.

Sphincter injection of botulinum toxin A (BoNT-A) was first used to treat detrusor sphincter dyssynergia following spinal injury when inappropriately timed but qualitatively normal EMG activity occurs in the sphincter with detrusor contraction. However some recent publications have reported a restoration of detrusor function after sphincter injections of botulinum toxin A in women with non-neurological conditions, although insufficient detail is given in those papers to know if the patients had FS. Although, Fowler used sphincter botulinum toxin injections 15 years ago in an attempt to treat that condition it was concluded then that the intervention was not effective. This was possibly because a much lower dose was used compared with the recently reported successful studies, in which 100 U Botox® were used.

Objectives: The aim of this small scale, open label pilot study is to obtain data about the response of women with a definite diagnosis of FS after an injection of 100 U Botox® (BoNT-A) into the striated urethral sphincter. If there is evidence for a positive response the data will form the basis for a future large scale, placebo controlled, grant funded study.

Method: 5 women with complete urinary retention due to the abnormality of sphincter relaxation demonstrated to be characteristic of FS and 5 women with the same sphincter abnormality but with obstructed voiding will be fully studied to document the severity and extent of their sphincter-bladder dysfunction.

Pre-treatment assessment will include the standard investigations appropriate for women with complete urinary retention or obstructed voiding which have been shown to be characteristically abnormal in FS. These are urine flow rate (if voiding), cystometry, urethral pressure profile, sphincter volume. The definitive diagnosis rests on the findings of sphincter EMG and as this test is uncomfortable it will be possible to combine the necessary EMG recording with the injection of the Botox® if the patient consents to enter the study.

The injection treatment will be an outpatient procedure (estimated to take less than 15 minutes): following 1ml of 1% or 2% lignocaine injected either side of the urethral orifice, 100 U Botox® dissolved in 2mls of saline will be injected, 1ml on each side into the striated urethral sphincter under EMG control.

The effect of BoNT-A injected into other striated muscle is known to have an onset within 3-4 days and duration of action of 6 weeks. The patients will therefore be followed up at 1, 4, and 10 weeks following treatment with flowmetry and ultrasound residual volumes and IPSS questionnaire. The pre intervention investigations of cystometry, urine flow rate (if voiding) and residual volume measured by ultrasound, urethral pressure profile will be repeated at 4 weeks. Sphincter EMG will only be repeated in patients who have shown a highly significant response i.e. restoration of detrusor contraction in women who previously had complete urinary retention or elimination of post void residual volume in women with obstructed voiding.

Outcome measures Primary

* Improvement in urinary flow rates (as assessed by uroflowmetry and measured in mL/sec) by more than 50% after botulinum toxin compared to baseline in women with obstructed voiding
* Restoration of voiding (either yes or no) after botulinum toxin for women in complete urinary retention

Secondary

* Improvement of post void residual urine (as assessed by bladder scan and measured in mL) compared to baseline after botulinum toxin. A reduction to less than 100mls would be considered clinically significant.
* Improvement in lower urinary tract symptoms as assessed by an improvement in scores on the IPSS (International Prostate Symptom score) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old or over with diagnosed Fowler's syndrome and abnormal sphincter function i.e. raised UPP {MUCP>(92 - patient age in years) cmH2O} (Edwards and Malvern 1974), increased sphincter volume(if measured) (greater than 1.8 cm3) and if voiding, evidence of obstructed outflow. (Sphincter EMG will be recorded at the time of injection.)
* Willing to give written informed consent
* Willing to attend the necessary follow up visits
* On effective contraception if sexually active - oral contraceptive pill (>3 months use), condoms, intrauterine contraceptive device, depot injection

Exclusion Criteria:

* Previous urethral surgery (other than urethral dilatation)
* Neurological disease
* Pregnant or lactating women and those planning pregnancy
* Anticoagulant therapy at the time of inclusion*.
* On drugs that might interfere with neuromuscular transmission (e.g. aminoglycosides)
* Pain thought to originate from the urinary tract
* Unsuitable past medical history e.g. frequent epilepsy, uncontrolled hypertension, severe coronary artery disease.
* Symptomatic Urinary Tract Infection with a positive urine culture
* Participation in a clinical trial involving an investigational product in the last 3 months
* Patients who are unable to understand or speak English, as this is a pilot study involving very few patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Improvement in urinary flow rates as assessed by uroflowmetry by more than 50% | 10 weeks
  Improvement in urinary flow rates (as assessed by uroflowmetry and measured in mL/sec) by more than 50% after botulinum toxin compared to baseline in women with obstructed voiding
Restoration of voiding for women in complete urinary retention | 10 weeks
  Restoration of voiding (either yes or no) after botulinum toxin for women in complete urinary retention

SECONDARY OUTCOMES:
Improvement of post void residual urine compared to baseline | 10 weeks
  Improvement of post void residual urine (as assessed by bladder scan and measured in mL) compared to baseline after botulinum toxin. A reduction to less than 100mls would be considered clinically significant
Improvement in lower urinary tract symptoms as assessed by an improvement in scores on the IPSS questionnaire | 10 weeks
  Improvement in lower urinary tract symptoms as assessed by an improvement in scores on the IPSS (International Prostate Symptom score) questionnaire

REFERENCES:
- [Background] Dykstra DD, Sidi AA, Scott AB, Pagel JM, Goldish GD. Effects of botulinum A toxin on detrusor-sphincter dyssynergia in spinal cord injury patients. J Urol. 1988 May;139(5):919-22. doi: 10.1016/s0022-5347(17)42717-0. PMID 3361663
- [Result] Dasgupta R, Wiseman OJ, Kitchen N, Fowler CJ. Long-term results of sacral neuromodulation for women with urinary retention. BJU Int. 2004 Aug;94(3):335-7. doi: 10.1111/j.1464-410X.2004.04979.x. PMID 15291863
- [Result] Swinn MJ, Wiseman OJ, Lowe E, Fowler CJ. The cause and natural history of isolated urinary retention in young women. J Urol. 2002 Jan;167(1):151-6. PMID 11743295